CLINICAL TRIAL: NCT00000363
Title: Acute Otitis Media: Adjuvant Therapy to Improve Outcome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDCD-1160; R01DC002620-04 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2006-04-24 (Estimated); Status verified 2006-04

CONDITIONS: Otitis Media
Keywords: Antibiotics; Adrenal Cortex Hormones; Histamine H1 Antagonists; Infant; Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Histamine Antagonists; Adrenal Cortex Hormones

INTERVENTIONS:
Drug: Antihistamine
Drug: Corticosteroid

SUMMARY:
Acute otitis media is one of the most common diseases of childhood and is one of the major causes of hearing loss in children. Despite the availability of effective antibiotic therapy for otitis media, treatment failures, persistent effusions, and recurrences are common. This Phase III outpatient study aims to test whether adjuvant therapy (an antihistamine or a corticosteroid), in addition to antibiotic therapy, improves the acute and long-term outcomes of patients with acute otitis media. This study is targeted to recruiting 200 infants (age less than one year); patient (and parent) participation is estimated to continue for one year after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Have had two documented prior episodes of acute otitis media.
* Have no current middle ear effusion (fluid).

Exclusion Criteria:

* Have chronic otitis media.
* Have acute otitis media in addition to chronic otitis media.

Ages: 2 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Study Completion 2001-06

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tasnee Chonmaitree, Study Chair
Locations (1):
- Univ of Texas Med Branch Children's Hosp, Galveston, Texas, United States

REFERENCES:
- [Background] Chonmaitree T, Saeed K, Uchida T, Heikkinen T, Baldwin CD, Freeman DH Jr, McCormick DP. A randomized, placebo-controlled trial of the effect of antihistamine or corticosteroid treatment in acute otitis media. J Pediatr. 2003 Sep;143(3):377-85. doi: 10.1067/S0022-3476(03)00293-2. PMID 14517524
- [Background] McCormick DP, Saeed K, Uchida T, Baldwin CD, Deskin R, Lett-Brown MA, Heikkinen T, Chonmaitree T. Middle ear fluid histamine and leukotriene B4 in acute otitis media: effect of antihistamine or corticosteroid treatment. Int J Pediatr Otorhinolaryngol. 2003 Mar;67(3):221-30. doi: 10.1016/s0165-5876(02)00372-5. PMID 12633920